CLINICAL TRIAL: NCT05477628
Title: Nutrition Recommendation Intervention trialS in Children's Healthcare
Acronym: NuRISH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Toronto Public Health (Other Government); University of Toronto (Other); Unity Health Toronto (Other); Applied Health Research Centre (Other); McMaster University (Other); Pediatric Alliance of Ontario (Unknown); Canadian Paediatric Society (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Jonathon L Maguire, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 3606
Record Dates: First submitted 2022-06-02; First posted 2022-07-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Obesity, Childhood; Nutrition; Health Risk Behaviors; Breastfeeding; Exclusive Breastfeeding; Diabetes
Keywords: Lower adiposity; Higher breastfeeding self-efficacy; Higher centre-based childcare attendance; Improved child development and mental health; Lower cardiovascular risk factors; Better dietary quality; Lower healthcare and overall societal costs
MeSH Terms: conditions — Pediatric Obesity; Health Risk Behaviors; Breast Feeding; Diabetes Mellitus; Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This will be a pragmatic, randomized, longitudinal factorial Trials within Cohorts (TwiCs) clinical trial. This study will be a direct comparison of two HCP prescriptions provided randomly at the individual level: 1) Optimal breastfeeding with mobile lactation consultant support vs. usual care and 2) High-quality childcare starting at 1 year of age vs. usual care. We will combine TwiCs methods with a longitudinal factorial design to enhance the integration of cohort study and factorial trial designs.
Who Masked: Outcomes Assessor
Masking Description: To reduce the risk of bias, all research assistants who collect baseline and outcome data will be blinded. All other study personnel, including data analysts, will also be blinded to group allocation. Due to the nature of the intervention, children and parents cannot be blinded, but they will be blinded to trial hypotheses. Healthcare providers who provide the interventions also cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants who are randomized to the control group will receive usual care from their health care practitioners.
  Interventions: Other: Control Group
- Intervention Group (Experimental): Participants who are randomized to Intervention Group will receive one of three possible "scenarios": 1) Childcare Navigator Support, 2) Breastfeeding support via Lactation Consultant, 3) both Childcare Navigator Support and Breastfeeding support via Lactation.
  Interventions: Other: Childcare Navigator; Other: Lactation Consultant; Other: Lactation Consultant Support and Childcare Navigator Support

INTERVENTIONS:
Other: Childcare Navigator — Participants will be contacted by the CN to assist with access to centre-based childcare after enrolment. The CN will: a) educate the family on the benefits of centre based childcare; b) facilitate placement of the child on waiting lists for funding and centre based childcare placement in their neighbourhood with the aim of having full-time centre based childcare start at 1 year of age; and c) work with the family to overcome barriers to childcare placement prior to and during childcare. It is expected that the child will be in full-time centre-based childcare for a minimum of 12 months.
  Control: All children randomized to the control condition will receive age-appropriate nutritional recommendations as part of routine healthcare according to the Rourke Baby Record.
  Other Names: (CN)
  Arms: Intervention Group
Other: Lactation Consultant — Participants will be contacted by the LC on the same day as their first primary healthcare visit. They will also receive age-appropriate nutrition recommendations according to the Rourke Baby Record. The LC will be an International Board Certified Lactation Consultant (IBCLC) who will provide scheduled and on-call visits, along with phone calls, video conferencing, and text messaging as needed to support exclusive breastfeeding (using virtual care modalities as appropriate during COVID-19). The LC will contact the family once per week for the first 4 weeks to support breastfeeding technique and help with breastfeeding problems such as latching difficulties, painful nursing, and low milk production, monthly thereafter and provide on-call support as required to support exclusive breastfeeding through 6 months of age.
  Control: All children randomized to the control condition will receive age-appropriate nutritional recommendations as part of routine healthcare.
  Other Names: (LC)
  Arms: Intervention Group
Other: Lactation Consultant Support and Childcare Navigator Support — This intervention is a combination of the two interventions described above.
  Other Names: LC+CN
  Arms: Intervention Group
Other: Control Group — All children randomized to the control condition will receive age-appropriate nutritional recommendations as part of routine healthcare.
  Arms: Control Group

SUMMARY:
NuRISH is a suite of clinical trials for children from low-income families which will determine whether primary healthcare prescription for: 1) Optimal breastfeeding with support from a mobile lactation consultant vs. usual care and 2) High-quality childcare starting at 1 year vs. usual care can prevent childhood obesity, and improve cardiovascular, developmental and mental health at 2 years of age.

DETAILED DESCRIPTION:
Canada's children are falling behind. One in 4 are overweight or obese and more than 1 in 3 have factors that put them at risk for cardiovascular disease as adults. Children from low income families are 70% more likely to be overweight or obese. Research across disciplines has shown that early life nutrition has profound effects on childhood obesity, development, mental health, and lifetime success. Optimizing early life nutrition to reduce inequalities in childhood obesity and its consequences is a promising approach. Through this application, we will be using a longitudinal factorial design within an ongoing cohort study(TARGet Kids!). The longitudinal factorial design involves randomizing the same children to multiple interventions, providing the opportunity to evaluate the effect of individual interventions as well as the multiplicative effects of a combination of interventions over time. This design increases the feasibility and lowers the cost relative to conducting 2 separate trials. This will be a pragmatic, randomized, longitudinal factorial Trials within Cohorts (TwiCs) clinical trial. This study will be a direct comparison of two primary healthcare interventions provided randomly at the individual level: 1) Lactation Consultant (LC) support vs. usual care; 2) Childcare Navigator (CN) support vs. usual care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy by parental report
* <32 weeks gestation
* 0-1 week of age
* First birth /first time parents

Exclusion Criteria:

* Children with a syndrome associated with obesity or developmental delay

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 620 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
zBMI | 2-year primary healthcare visit
  The primary outcome measure will be age and sex standardized BMI z-score (zBMI), which will be measured at the 2-year primary healthcare visit. zBMI is an important outcome that is predictive of adiposity in later childhood, adolescence and adulthood. Data including birthweight and length, and repeated measures of weight and length will be used to calculate zBMI growth trajectories.

SECONDARY OUTCOMES:
breastfeeding self-efficacy | 6 months
  change in breastfeeding self-efficacy measured by lactation consultant logs
exclusive breastfeeding duration | 6 months
  change in exclusive breastfeeding duration
Childcare attendance | 2 years of age
  change in centre-based childcare attendance measured by attendance logs
cognitive development | 2 years of age
  To capture child's development, the Ages and Stages Questionnaire will be administered. The Ages and Stages Questionnaire identifies infants, toddlers and preschool aged children at risk of a developmental delay in five developmental domains: Communication, Gross Motor, Fine Motor, Problem Solving and Personal Social Behaviour. Each domain consists of six questions about important age-specific developmental milestones. If a child scores between 1 and 2 below the normative mean on any domain, rescreening is recommended. When a child scores 1 below the normative mean on two or more domains, or 2 below the normative mean on at least one domain, a referral to a health care professional is recommended.
maternal mental health | 2 years of age
  change in maternal mental health, measured by the Edinburgh Postnatal Depression Scale at 2 years of age. The scale was developed for screening postpartum women in outpatient, home visiting settings, or at the 6 -8 week postpartum examination. Consisting of 10 questions, each response is scored 0, 1, 2, or 3 according to increased severity of the symptom. Items marked with an asterisk (*) are reverse scored (i.e., 3, 2, 1, and 0). The total score is determined by adding together the scores for each of the 10 items. A woman scoring 9 or more points or indicating any suicidal ideation - that is she scores 1 or higher on question #10 - should be referred immediately for follow-up. Even if a woman scores less than 9, if the clinician feels the client is suffering from depression, an appropriate referral should be made.
mental health | 2 years of age
  Child's mental health captured by the Strengths and Difficulties Questionnaire. The questionnaire consists of 25 items subdivided into four difficulties scales, emotional symptoms, conduct problems, inattention-hyperactivity and peer problems, and a separate fifth strength scale, prosocial behavior. All subscales have five questions. Each item has to be scored on a 3-point scale with 0 = 'not true', 1 = 'somewhat true' and 2 = 'certainly true'. A higher score indicates more emotional and behavioral problems.
blood pressure | 2 years of age
  change in cardiovascular risk factors for the child
non-HDL | 2 years of age
  change in cardiovascular risk factors for the child
LDL | 2 years of age
  change in cardiovascular risk factors for the child
triglyceride | 2 years of age
  change in cardiovascular risk factors for the child
HDL | 2 years of age
  change in cardiovascular risk factors for the child
TC | 2 years of age
  change in cardiovascular risk factors for the child
glucose | 2 years of age
  change in cardiovascular risk factors for the child
hsCRP | 2 years of age
  change in cardiovascular risk factors for the child
HbA1C | 2 years of age
  change in cardiovascular risk factors for the child
Dietary Quality | 2 years of age
  total caloric intake captured through the Automated Self-Administered 24-hour Dietary Assessment Tool of the child and mother at 2 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Maguire, MD,FRCPC,MSc, Principal Investigator — The Hospital for Sick Children

IPD SHARING:
Plan to Share IPD: No